CLINICAL TRIAL: NCT01235533
Title: The Assessment for the Effects of Health Products on Depression and Cognitive Function:Fish Oil in Patients With Late-life Depression
Brief Title: Fish Oil Supplementation in Late-life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Psychiatric Center, Taiwan (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: CHIH-CHIANG CHIU, Taipei City Psychiatric Center, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 95004-62-161
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Late-Life Depression
Keywords: late-life depression; recurrence of depression; cognition; N-3 polyunsaturated fatty acids
MeSH Terms: interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-3 fatty acids (Experimental): Participants in this arm were received three capsules of n-3 fatty acids. Each capsule included 600mg eicosapentanoic acid (20:5n-3), 400 mg of docosahexanoic acid (22:6n-3), tertiary-butylhydroquinone 0.2 mg/g and tocopherols 2 mg/g。
  Interventions: Dietary Supplement: N-3 polyunsaturated fatty acids
- Placebo (Placebo Comparator): Participants in this arm were received three identical capsules per day. All capsules included olive oil.
  Interventions: Dietary Supplement: N-3 polyunsaturated fatty acids

INTERVENTIONS:
Dietary Supplement: N-3 polyunsaturated fatty acids — Three capsules per day. Each capsule included 600mg eicosapentanoic acid (20:5n-3), 400 mg of docosahexanoic acid (22:6n-3), tertiary-butylhydroquinone 0.2 mg/g and tocopherols 2 mg/g.
  Other Names: Fish oil

SUMMARY:
To investigate whether fish oil supplementation, compared to placebo (olive oil), could have better effects on depression course and cognitive function in older people with major depression.

DETAILED DESCRIPTION:
Patients with late-life depression were reported cognitive impairment, especially in information-processing speed, working memory, attention and episodic memory, even after depressive symptoms subside and some of them further progress to dementia in two to four years. Several epidemiological studies, fatty acid comparison studies, animal studies, and clinical trials found that omega-3 polyunsaturated fatty acids (PUFAs) were significantly associated with the major depression, cognitive decline in general population and Alzheimer's disease. Until now, there is no study investigating the effects of n-3 PUFAs on depressive symptoms and cognition in patients with late-life depression. Thus, the aims of this study were to investigate whether fish oil supplementation, compared to placebo (olive oil), could have better effects on depression course and cognitive function in older people with major depression.

ELIGIBILITY:
Inclusion Criteria:

* An age range of 60 years old or over;
* A previous diagnosis of major depressive disorder according to the Chinese version of Structured Clinical Interview for DSM IV-TR Axis-I Disorder;
* Depressive symptoms were stable for at least three consecutive weeks and the 17-item Hamilton Depression Rating Scale score less or equal to 10.
* Capacity to provide informed consent.

Exclusion Criteria:

* People with severe or acute medical illness ( such as metastatic cancer, brain tumor, decompensated cardiac, hepatic, or renal failure, or myocardial infarction or stroke) within the 3 months preceding the study.
* Those who had neurological disorders involving central nervous system, such as delirium, Parkinson's disease, aphasia or multiple sclerosis)
* Prominent cognitive impairment, defined as the Chinese version of Mini-Mental State examination score less than 17.
* People with alcoholism, defined by a score of 8 or higher in male and of 6 or higher in female on the Chinese version of the Alcohol Use Disorders Identification Test (AUDIT) questionnaire.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Recurrence of depression | week 8, 16, 24, 32, 40, 48
  Definition of recurrence of depression (between last visit and current visit):
  1. Fulfilled diagnosis of major depressive episode according to DSM-IV-TR
  2. Score of sucide subscale in 17-item Hamilton Depression Rating was 3 or over
  3. Hospitalization due to depression

SECONDARY OUTCOMES:
Change of cognitive function | Week 48
  Comparison of cognitive function at week 48 between two groups after adjustment for age, gender, education and baseline cognitive funciton

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-CHIANG CHIU, M.D., Principal Investigator — Department of Psychiatry, Taipei City Psychiatric Center, Taipei City Hospital
Locations (2):
- Taiwan (2):
  - Chih-Chiang Chiu, Taipei
  - Department of Psychiatry, Cathay General Hospital, Taipei

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851